CLINICAL TRIAL: NCT05015712
Title: Effects of Moderate Intensity Continuous Training (MICT) on Cardiopulmonary Function in Patients After Transcatheter Aortic Valve Implantation (TAVI): A Randomized Controlled Trial
Brief Title: Effects of MICT on Cardiopulmonary Function in Patients After TAVI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Han Yaling, MD (Other)
Responsible Party: Sponsor-Investigator, Han Yaling, MD, Director of Department of Cardiology, Principal Investigator, Shenyang Northern Hospital
Organization: Shenyang Northern Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: N2021-08
Record Dates: First submitted 2021-08-07; First posted 2021-08-20 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Valve Disease, Aortic; Cardiac Rehabilitation
Keywords: transcatheter aortic valve implantation; cardiac rehabilitation; cardiopulmonary function
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- moderate intensity continuous training (Experimental)
  Interventions: Behavioral: moderate intensity continuous training
- guideline control (No Intervention): Patients assigned to the guideline control just received 1-time advice on training according to guidelines.

INTERVENTIONS:
Behavioral: moderate intensity continuous training — Moderate intensity continuous training was scheduled 3 times per week for 3 months. Every sessions included warm-up (<50% target intensity for 2 min then gradually increasing load 1-10 W/min up to 100% target intensity for 5-10 min), exercise phase (100% target intensity (heart rate at anaerobic threshold±5) starting with 20 min and gradually lengthening up to 45 min in the 1 month as well as 45 min in another 2 months), cool down with gradual reduction of load within 3 min. The target intensity will be determined by the heart rate at anaerobic threshold measured by cardiopulmonary exercise test (CPET). The intensity will be adjusted after implementation of CPET and will keep at a minimum intensity, gradually increasing to the maximum intensity every month. Moreover, patients will be instructed to complete 2 supervised sessions and 1 home-based session during the 1 month and then to continue 3 home-based session for a further 2 months.
  Arms: moderate intensity continuous training

SUMMARY:
Cardiac rehabilitation (CR), particularly regular exercise, can improve the cardiopulmonary function, exercise capacity, and quality of life for patients undergoing transcatheter aortic valve implantation (TAVI). Consequently, the patients after TAVI will be enrolled in our randomized controlled trial to demonstrate if the moderate-intensity continuous training (MICT) can improve the cardiopulmonary function compared with the control group after receiving treatment for 12 weeks. Moreover, we will provide new insights regarding whether cardiac systolic function or cardiac diastolic function is mainly improved after regular exercise for TAVI patients. As a result, the principal hypothesis of our study is that MICT will improve the cardiopulmonary function and can extremely affect the cardiac diastolic function of patients with TAVI after the implementation of exercise for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* TAVI after 1 month
* able to start cardiac rehabilitation(CR) as judged by the study investigators
* age >18 years old
* 6-min walk distance (6MWD) ≥100m
* patients able to provide the informed consent before randomization

Exclusion Criteria:

* exercise-limiting comorbidities such as primarily orthopedic, neurological conditions that would exclude the patients from participating in CR
* linguistic deficits
* patient unwilling or unable to provide written informed consent
* patients with acute systemic diseases e.g. hyperthyroidism, electrolyte disturbances, uncontrolled diabetes, hemoglobin< 9 g/dL, uncontrolled asthma, severe obstructive pulmonary disease (forced expiratory volume in 1 second<50%), respiratory failure, and pulmonary embolism
* echocardiographic signs of prosthesis dysfunction including valve orifice area of <1.2 cm2 plus a mean transaortic pressure gradient of ≥20 mmHg, or a velocity of ≥3 m/s, at least moderate paravalvular regurgitation, signs of ischemia, severe arrhythmias, or hemodynamic deterioration during the exercise test
* decompensated heart failure (New York Heart Association (NYHA) class IV)
* patients with irreversible atrial or ventricular arrhythmias or patients with severe atrioventricular block
* bradycardia (heart rate<60bpm) or patients who need implantation of a pacemaker or implantable cardioverter defibrillators (ICD)
* recent history of sudden cardiac death syndrome
* suspected aortic dissection, pericarditis, hypertrophic obstructive cardiomyopathy and subacute bacterial endocarditis
* untreated or uncontrolled hypertension (systolic blood pressure > 180 mmHg and/or diastolic blood pressure >110 mmHg) or hypotension (systolic blood pressure <90 mmHg and/or diastolic blood pressure <60mmHg)
* cerebral hemorrhage, subarachnoid hemorrhage, cerebral thrombosis, cerebral embolism or other brain disease history
* active or recent major bleeding or bleeding predisposition
* coronary artery bypass grafting (CABG) within 3 months
* renal insufficiency (serum creatinine >2.5 mg/dl)
* planning to, or participation in another intervention study within 3 months
* patients with exercise intolerance or poor exercise endurance
* patients who are currently receiving systematic training
* researchers think it is not suitable to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-08-20 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
change in peak oxygen uptake (peak VO2) after 3 months | 3 months and 1 year

SECONDARY OUTCOMES:
6-min walk distance | 3 months and 1 year
the Medical Outcomes Study 12-Item Short-Form Health Survey (SF-12) | 3 months and 1 year
New York Heart Association class (NYHA) | 3 months and 1 year
  The NYHA is measured by Classification of NYHA heart function
E/e' | 3 months and 1 year
  it is measured by echocardiography
E/A | 3 months and 1 year
  it is measured by echocardiography
left atrial volume index(LAVI) | 3 months and 1 year
  it is measured by echocardiography
left ventricular ejection fraction(LV-EF) | 3 months and 1 year
  it is measured by echocardiography
mean pressure gradient(PGmean) | 3 months and 1 year
  it is measured by echocardiography
maximal pressure gradient (PGmax) | 3 months and 1 year
  it is measured by echocardiography
maximal velocity(Vmax) | 3 months and 1 year
  it is measured by echocardiography
valve orifice area | 3 months and 1 year
  it is measured by echocardiography
N-terminal pro-brain natriuretic peptide (NT-proBNP) | 3 months and 1 year
C-reactive protein(CRP) | 3 months and 1 year
hemoglobin | 3 months and 1 year
cholesterol | 3 months and 1 year
triglyceride | 3 months and 1 year
high density lipoprotein (HDL) | 3 months and 1 year
low density lipoprotein (LDL) | 3 months and 1 year
Major adverse cardiovascular events | 3 months and 1 year
  Major adverse cardiovascular events is a composite endpoint of death, stroke, revascularization, and myocardial infarction.
change in peak oxygen uptake (peak VO2) after 1 year | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Ling Han, PhD, Principal Investigator — Department of Cardiology, General Hospital of Northern Theater Command, Shenyang 110016, China
Locations (1):
- Ya-Ling Han, Shenyang, Liaoning, China